CLINICAL TRIAL: NCT02430870
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability, and Pharmacokinetic Study of Escalating Multiple Oral TAK-648 Doses in Healthy Japanese Subjects and Subjects With Type 2 Diabetes Mellitus
Brief Title: TAK-648 Multiple-Rising Dose Study in Healthy Japanese Participants and Non-Japanese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-648-1002; U1111-1165-3437 (Registry Identifier: WHO)
Record Dates: First submitted 2015-04-24; First posted 2015-04-30 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part 1 Cohort 1: TAK-648 0.35 mg (Experimental): Participants with T2DM on a stable dose of metformin in study Part 1, Cohort 1 received TAK-648 0.35 mg, solution, orally, single dose on Day 1, no drug administration on Days 2 to 3, followed by once daily (QD) doses starting on Day 4 and continuing through Day 17 (14 days).
  Interventions: Drug: TAK-648
- Part 1 Cohort 2: TAK-648 0.80 mg (Experimental): Participants with T2DM on a stable dose of metformin in study Part 1, Cohort 2 received TAK-648 0.80 mg, solution, orally, single dose on Day 1, no drug administration on Days 2 to 3, followed by once daily (QD) doses starting on Day 4 and continuing through Day 17 (14 days).
  Interventions: Drug: TAK-648
- Part 1: Placebo Cohort 1-2 (Placebo Comparator): Participants with T2DM on a stable dose of metformin in study Part 1 received placebo-matching TAK-648, solution, orally, single dose on Day 1, no drug administration on Days 2 to 3, followed by once daily (QD) doses starting on Day 4 and continuing through Day 17 (14 days).
  Interventions: Drug: Placebo
- Part 2 Cohort 1: TAK-648 0.05 mg (Experimental): Healthy participants of Japanese descent in study Part 2, Cohort 1 received TAK-648 0.05 mg, solution , orally, single dose on Day 1, no drug administration on Days 2 to 3, followed by multiple QD doses starting on Day 4 and continuing through Day 10 (7 days).
  Interventions: Drug: TAK-648
- Part 2 Cohort 2: TAK-648 0.15 mg (Experimental): Healthy participants of Japanese descent in study Part 2, Cohort 2 received TAK-648 0.15 mg, solution, orally, single dose on Day 1, no drug administration on Days 2 to 3, followed by multiple QD doses starting on Day 4 and continuing through Day 10 (7 days).
  Interventions: Drug: TAK-648
- Part 2 Cohort 3: TAK-648 0.35 mg (Experimental): Healthy participants of Japanese descent in study Part 2, Cohort 3 received TAK-648 0.35 mg, solution, orally, single dose on Day 1, no drug administration on Days 2 to 3, followed by multiple QD doses starting on Day 4 and continuing through Day 10 (7 days).
  Interventions: Drug: TAK-648
- Part 2 Cohort 4: TAK-648 0.80 mg (Experimental): Healthy participants of Japanese descent in study Part 2, Cohort 4 received TAK-648 0.80 mg, solution, orally, single dose on Day 1, no drug administration on Days 2 to 3, followed by multiple QD doses starting on Day 4 and continuing through Day 10 (7 days).
  Interventions: Drug: TAK-648
- Part 2: Placebo Cohort 1-4 (Placebo Comparator): Healthy participants of Japanese descent in study Part 2, received TAK-648 placebo-matching solution, orally, single dose on Day 1, no drug administration on Days 2 to 3, followed by multiple QD doses starting on Day 4 and continuing through Day 10 (7 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-648 — TAK-648 solution
  Arms: Part 1 Cohort 1: TAK-648 0.35 mg; Part 1 Cohort 2: TAK-648 0.80 mg; Part 2 Cohort 1: TAK-648 0.05 mg; Part 2 Cohort 2: TAK-648 0.15 mg; Part 2 Cohort 3: TAK-648 0.35 mg; Part 2 Cohort 4: TAK-648 0.80 mg
Drug: Placebo — TAK-648 placebo-matching solution
  Arms: Part 1: Placebo Cohort 1-2; Part 2: Placebo Cohort 1-4

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled, 2-center, multiple-dose study in healthy participants and participants with type 2 diabetes mellitus (T2DM). This study will evaluate the safety, tolerability and pharmacokinetics (PK) of TAK-648 when administered as multiple oral doses of TAK-648 solution at escalating dose levels in healthy participants of Japanese decent and participants with T2DM.

DETAILED DESCRIPTION:
The drug being evaluated in this study is TAK-648 for the treatment of T2DM.

This study will consist of 2 parts: (1) multiple ascending doses in participants with T2DM treated with a stable dose of metformin, (2) multiple ascending doses in healthy participants of Japanese descent.

Part 1 of this study will consist of 2 multiple dose treatment cohorts (Cohorts 1-2 designated as P1C1 and P1C2) dosed sequentially in escalating order. The projected doses of TAK-648 for Part 1 are 0.15 and 0.35 mg of TAK-648, but may be adjusted higher or lower, and additional cohorts may be added, based on available safety and pharmacokinetic (PK) data. All cohorts in Part 1 will consist of 8 (2 placebo) T2DM participants.

Part 2 of this study will consist of 3 multiple dose treatment cohorts (Cohorts 1-3 designated as P2C1, P2C2 and P2C3) in healthy participants of Japanese descent dosed sequentially in escalating order. The projected doses of TAK-648 chosen for Part 2 are 0.05, 0.15 and 0.35 mg of TAK-648, but may be adjusted higher or lower based on available safety and PK data. All cohorts in Part 2 will consist of 8 (2 placebo) healthy participants of Japanese descent.

Additional cohorts may be recruited and studied as necessary to better evaluate safety, tolerability, PK, and/or PD parameters.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

1. Is an adult male or female and has a historical diagnosis of type 2 diabetes mellitus (T2DM) disease.
2. Is aged 18 to 65 years, inclusive, at the time of informed consent and first study medication dose.
3. Weighs at least 55 kg and has a body mass index (BMI) ≥23.0 kg/m^2 and ≤35.0 kg/m^2 at Screening.
4. Has a systolic blood pressure >90 and ≤150 mm Hg and a diastolic blood pressure of >60 and ≤90 mm Hg at Screening and at Check-in (Day -2). If out of range, may be repeated once for eligibility determination within a maximum of5 minutes.
5. Has a calculated creatinine clearance >60 mL/min at Screening and Check-in (Day -2).
6. Has been treated for inadequate glycemic control with a stable dose of metformin for the least 8 weeks prior to Screening.
7. Has a glycosylated hemoglobin (HbA1c) level between 6.5% and 10.0%, inclusive at Check-in (Day -2).
8. Has a fasting C-peptide concentration ≥0.8 ng/mL at Screening.
9. Has no medical history of type 1 diabetes mellitus (T1DM), hypoglycemia unawareness, diabetic ketoacidosis or hyperosmolar coma.

Part 2:

1. Is a healthy adult male or female of Japanese descent (born to Japanese parents and grandparents) and have lived outside of Japan for less than 5 years, inclusive.
2. Is aged 20 to 55 years, inclusive, at the time of informed consent and first study medication dose.
3. Weighs at least 45 kg and has a BMI from 17.0 to 25.0 kg/m^2, inclusive at Screening.
4. Has a systolic blood pressure >90 and ≤150 mm Hg and a diastolic blood pressure of >60 and ≤90 mm Hg at Screening and at Check-in (Day -2). If out of range, may be repeated once for eligibility determination within a maximum of 5 minutes.
5. Has a calculated creatinine clearance >60 mL/min at Screening and Check-in (Day -2).

Exclusion Criteria:

Part 1:

1. Has Screening or Check-in (Day -2) laboratory values of serum creatinine ≥1.5 mg/dL for males or ≥1.4 mg/dL [females] or abnormal creatinine clearance.
2. Has a history of T1DM, hypoglycemia unawareness, diabetic ketoacidosis, or hyperosmolar coma.
3. Has a history of any clinically significant retinopathy, which is defined as more than moderate nonproliferative diabetic retinopathy or any stage of proliferative diabetic retinopathy or any history of laser-treated retinopathy.
4. Has received any antihyperglycemic medication with the exception of metformin within the previous 12 weeks of Check-in (Day -2) or the subject has changed the dose of metformin within the previous 8 weeks of Screening.
5. Is expecting to receive, receiving or has received systemic glucocorticoid therapy for a duration longer than 5 days within the previous 12 weeks of Check-in (Day -2).

Parts 1 and 2:

1. Has received any investigational compound within 30 days prior to the first dose of study medication.
2. Has received TAK-648 in a previous clinical study or as a therapeutic agent.
3. Has any significant medical histories or currently uncontrolled clinical conditions, which may not be safe for participants to participate in the study, may impact the ability of the participant to participate in the study, or may potentially confound the study results. The concerned significant medical histories and uncontrolled clinical conditions include (may not be limited to) cardiovascular (such as ischemic heart disease, heart failure, cardiomyopathy, clinically significant arrhythmia, uncontrolled or unstable blood pressure), central nervous system, hepatic or hematopoietic disease(s), renal dysfunction, metabolic or endocrine dysfunction, pulmonary diseases including serious allergy and asthma hypoxemia, seizures, or allergic skin rash.
4. Has a history of significant GI disorders manifested with persistent, chronic or intermittent nausea, vomiting or diarrhea, or has a current or recent (within 6 months) GI disease that would influence the absorption of drugs (eg, a history or malabsorption, severe esophageal reflux, peptic ulcer disease or erosive esophagitis with frequent [more than once per week] occurrence of heartburn).
5. Has diagnosis of major depression, bipolar disorder or anxiety disorders, or has a risk of anxiety, depression, or insomnia according to the investigator's clinical judgment per HAM-D17 at Screening or has received any medication to treat any psychological disorders within 1 year.
6. Has a risk of suicide according to the investigator's clinical judgment per C-SSRS at Screening or has made a suicide attempt in the past 6 months prior to Screening.
7. Has a known hypersensitivity to any component of the formulation ofTAK-648, or to a PDE4 inhibitor (eg, roflumilast) or Listerine strips.
8. Has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -2).
9. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
10. Has taken any excluded medication, supplements, or food products.
11. If female, is pregnant or lactating or intending to become pregnant before, during, or within 12 weeks after participating in this study; or intending to donate ova during such time period.
12. If male, intends to donate sperm during the course of this study or for 12 weeks thereafter.
13. Has a history of cancer, except basal cell carcinoma that has been in remission for at least 5 years prior to Day 1.
14. Has a positive test result for HBsAg, anti-HCV, at Screening or a known history of human immunodeficiency virus infection.
15. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 6 weeks prior to Check-in (Day -2). Cotinine test is positive at Screening or Check-in (Day -2).
16. Has poor peripheral venous access.
17. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 30 days prior to Day 1.
18. Has a Screening or Check-in (Day -2) abnormal (clinically significant) ECG, including but not limited to those with evidence of prolonged QT/QTc interval at Baseline (eg, QTc interval >450 milliseconds) or those at risk for QT prolongation (eg with a family history of long QT syndrome). Entry of any subject with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator or medically qualified subinvestigator.
19. Has abnormal Screening or Check-in (Day -2) laboratory values that suggest a clinically significant underlying disease or participant with the following laboratory abnormalities: ALT and/or AST >2.5×ULN.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Anaheim, California
  - Chula Vista, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 02 April 2015 to 04 November 2015.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitus (T2DM) were enrolled in 1 of 3 treatment groups: placebo, 0.35 mg or 0.80 mg TAK-648 in Part 1. Healthy Japanese volunteers were enrolled in 1 of 5 treatment groups: placebo, 0.05 mg, 0.15 mg, 0.35 mg or 0.80 mg TAK-648 in Part 2.
Groups:
- Part 1 Cohort 1: TAK-648 0.35 mg: Participants with T2DM in study Part 1, Cohort 1 received TAK-648 0.35 mg, solution, orally, single dose on Day 1, no drug administration on Days 2 to 3, followed by once daily (QD) doses starting on Day 4 and continuing through Day 17 (14 days).
- Part 1 Cohort 2: TAK-648 0.80 mg: Participants with T2DM in study Part 1, Cohort 2 received TAK-648 0.80 mg, solution, orally, single dose on Day 1, no drug administration on Days 2 to 3, followed by once daily (QD) doses starting on Day 4 and continuing through Day 17 (14 days).
- Part 1: Placebo Cohort 1-2: Participants with T2DM in study Part 1 received placebo-matching TAK-648, solution, orally, single dose on Day 1, no drug administration on Days 2 to 3, followed by once daily (QD) doses starting on Day 4 and continuing through Day 17 (14 days).
Period: Part 1
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg | Part 1: Placebo Cohort 1-2 | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg | Part 2: Placebo Cohort 1-4
Started | 6 | 6 | 4 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 4 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg | Part 1: Placebo Cohort 1-2 | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg | Part 2: Placebo Cohort 1-4
Started | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 8
Completed | 0 | 0 | 0 | 6 | 6 | 6 | 5 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Voluntary Withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg | Part 1: Placebo Cohort 1-2 | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg | Part 2: Placebo Cohort 1-4 | Total
Number analyzed (Participants) | 6 | 6 | 4 | 6 | 6 | 6 | 6 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — Data presented for study Part 1 only. Age data for study Part 2 is reported in a separate baseline measure.
  years | 55.3 (8.04) [46 to 64] | 55.0 (7.01) [46 to 64] | 54.5 (7.77) [43 to 60] | NA (NA) [26 to 51] — Reported in a separate baseline measure. | NA (NA) [26 to 54] — Reported in a separate baseline measure. | NA (NA) [21 to 54] — Reported in a separate baseline measure. | NA (NA) [30 to 41] — Reported in a separate baseline measure. | NA (NA) [21 to 53] — Reported in a separate baseline measure. | 55.0 (7.08) [21 to 64]
Age, Continuous [Mean (Standard Deviation); unit: years] — Data presented for study Part 2 only. Age data for study Part 1 is reported in a separate baseline measure.
  years | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | 37.3 (9.63) | 36.0 (10.45) | 32.2 (12.48) | 33.0 (4.10) | 35.3 (9.82) | 34.8 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants] — Data presented for study Part 1 only. Gender data for study Part 2 is reported in a separate baseline measure.
  Participants
    Female | 0 | 3 | 4 | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | 6 | 3 | 0 | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants] — Data presented for study Part 2 only. Gender data for study Part 1 is reported in a separate baseline measure.
  Participants
    Female | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | 1 | 3 | 3 | 3 | 5 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | 5 | 3 | 3 | 3 | 3 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Number; unit: participants] — Data presented for study Part 1 only. Ethnicity data for study Part 2 is reported in a separate baseline measure.
  participants
    Hispanic or Latino | 6 (4.09) [165 to 176] | 5 (9.95) [155 to 179] | 4 (8.70) [147 to 163] | NA (NA) [NA to NA] — Reported in a separate baseline measure. | NA (NA) [NA to NA] — Reported in a separate baseline measure. | NA (NA) [NA to NA] — Reported in a separate baseline measure. | NA (NA) [NA to NA] — Reported in a separate baseline measure. | NA (NA) [NA to NA] — Reported in a separate baseline measure. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Non-Hispanic and Latino | 0 | 1 | 0 | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Number; unit: participants] — Data presented for study Part 2 only. Ethnicity data for study Part 1 is reported in a separate baseline measure.
  participants
    Non-Hispanic and Latino | NA (5.082) [83.3 to 98.6] — Reported in a separate baseline measure. | NA (17.359) [56.4 to 94.6] — Reported in a separate baseline measure. | NA (17.068) [54.0 to 89.5] — Reported in a separate baseline measure. | 6 (NA) [55.0 to 77.5] | 6 (NA) [49.4 to 77.7] | 6 (NA) [47.9 to 65.2] | 6 (NA) [52.4 to 81.3] | 8 (NA) [46.8 to 77.7] | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Number; unit: participants] — Data presented for study Part 1 only. Race data for study Part 2 is reported in a separate baseline measure.
  participants
    White | 6 (2.176) [27.2 to 33.9] | 6 (4.599) [22.9 to 34.4] | 4 (4.146) [24.3 to 33.7] | NA (NA) [19.5 to 24.9] — Reported in a separate baseline measure. | NA (NA) [20.3 to 25.1] — Reported in a separate baseline measure. | NA (NA) [18.7 to 23.8] — Reported in a separate baseline measure. | NA (NA) [20.2 to 26.3] — Reported in a separate baseline measure. | NA (NA) [19.0 to 24.8] — Reported in a separate baseline measure. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Number; unit: participants] — Data presented for study Part 2 only. Race data for study Part 1 is reported in a separate baseline measure.
  participants
    Asian | NA (534.56) — Reported in a separate baseline measure. | NA (709.93) — Reported in a separate baseline measure. | NA (645.98) — Reported in a separate baseline measure. | 6 (NA) | 6 (NA) | 6 (NA) | 6 (NA) | 8 (NA) | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants] — Data presented for study Part 1 only. Region of enrollment data for study Part 2 is reported in a separate baseline measure.
  participants
    United States | 6 | 6 | 4 | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Reported in a separate baseline measure. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants] — Data presented for study Part 2 only. Region of enrollment data for study Part 1 is reported in a separate baseline measure.
  participants
    United States | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | 6 (9.63) | 6 (10.45) | 6 (12.48) | 6 (4.10) | 8 (9.82) | NA — Total not calculated because data are not available (NA) in one or more arms.
Height [Mean (Standard Deviation); unit: cm] — Data presented for study Part 1 only. Height data for study Part 2 is reported in a separate baseline measure.
  cm | 171.5 (4.09) | 166.3 (9.95) | 155.5 (8.70) | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | 165.6 (9.75)
Height [Mean (Standard Deviation); unit: cm] — Data presented for study Part 2 only. Height data for study Part 1 is reported in a separate baseline measure.
  cm | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | 172.7 (5.32) | 169.0 (13.02) | 164.5 (6.57) | 166.3 (8.19) | 164.9 (8.43) | 167.3 (8.66)
Weight [Mean (Standard Deviation); unit: kg] — Data presented for study Part 1 only. Weight data for study Part 2 is reported in a separate baseline measure.
  kg | 91.45 (5.082) | 81.22 (17.359) | 73.38 (17.068) | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | 83.09 (14.895)
Weight [Mean (Standard Deviation); unit: kg] — Data presented for study Part 2 only. Weight data for study Part 1 is reported in a separate baseline measure.
  kg | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | 67.52 (9.055) | 65.40 (12.236) | 57.82 (6.421) | 64.47 (11.585) | 58.40 (10.206) | 62.45 (10.248)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Data presented for study Part 1 only. BMI data for study Part 2 is reported in a separate baseline measure.
  kg/m^2 | 31.12 (2.176) | 29.12 (4.599) | 30.00 (4.146) | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | 30.09 (3.587)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Data presented for study Part 2 only. BMI data for study Part 1 is reported in a separate baseline measure.
  kg/m^2 | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | NA (NA) — Reported in a separate baseline measure. | 22.58 (2.207) | 22.70 (1.531) | 21.33 (1.983) | 23.13 (2.234) | 21.34 (2.215) | 22.16 (2.072)
Metformin Dose [Mean (Standard Deviation); unit: mg] — Applies only to Part 1 only, participants with T2DM.
  mg | 1425.0 (534.56) | 1400.0 (709.93) | 1812.5 (645.98) | NA (NA) — Not Applicable: Healthy Participant | NA (NA) — Not Applicable: Healthy Participant | NA (NA) — Not Applicable: Healthy Participant | NA (NA) — Not Applicable: Healthy Participant | NA (NA) — Not Applicable: Healthy Participant | 1512.5 (615.49)
Duration of Type 2 Diabetes Mellitus (T2DM) [Mean (Standard Deviation); unit: years] — Applies only to Part 1 only, participants with T2DM.
  years | 12.7 (5.68) | 9.3 (5.16) | 9.0 (3.37) | NA (NA) — Not Applicable: Healthy Participant | NA (NA) — Not Applicable: Healthy Participant | NA (NA) — Not Applicable: Healthy Participant | NA (NA) — Not Applicable: Healthy Participant | NA (NA) — Not Applicable: Healthy Participant | 10.5 (4.99)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have at Least 1 Treatment-Emergent Adverse Event (TEAE) for Part 1
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to Day 34
Population: Safety Analysis Set included of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg | Part 1: Placebo Cohort 1-2
Number analyzed (Participants) | 6 | 6 | 4
percentage of participants | 83.3 | 33.3 | 100.0

2. Primary Outcome: Percentage of Participants Who Have at Least 1 Treatment-Emergent Adverse Event (TEAE) for Part 2
Description: as for outcome 1
Time Frame: Up to Day 26
Population: Safety Analysis Set included of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg | Part 2: Placebo Cohort 1-4
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
percentage of participants | 100.0 | 33.3 | 66.7 | 83.3 | 37.5

3. Primary Outcome: Percentage of Participants With Markedly Abnormal Laboratory Values at Least Once Post-dose During Dosing for Part 1
Time Frame: Up to Day 20
Population: Safety Analysis Set included of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg | Part 1: Placebo Cohort 1-2
Number analyzed (Participants) | 6 | 6 | 4
percentage of participants | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants With Markedly Abnormal Laboratory Values at Least Once Post-dose During Dosing for Part 2
Time Frame: Up to Day 13
Population: Safety Analysis Set included of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg | Part 2: Placebo Cohort 1-4
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
percentage of participants | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Percentage of Participants With Markedly Abnormal Vital Sign Values at Least Once Post-dose During Dosing for Part 1
Description: Vital signs included body temperature (oral), sitting blood pressure (after 5 minutes resting), respiration rate and pulse (bpm).
Time Frame: Up to Day 20
Population: Safety Analysis Set included of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg | Part 1: Placebo Cohort 1-2
Number analyzed (Participants) | 6 | 6 | 4
percentage of participants
  < Lower Criteria | 0 | 16.7 | 50.0
  > Upper Criteria | 16.7 | 0 | 0

6. Primary Outcome: Percentage of Participants With Markedly Abnormal Vital Sign Values at Least Once Post-dose During Dosing for Part 2
Description: Vital signs included body temperature (oral), sitting blood pressure (after 5 minutes resting), respiration rate and pulse (bpm),
Time Frame: Up to Day 13
Population: Safety Analysis Set included of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg | Part 2: Placebo Cohort 1-4
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
percentage of participants
  < Lower Criteria | 50.0 | 50.0 | 33.3 | 33.3 | 37.5
  > Upper Criteria | 0 | 16.7 | 0 | 0 | 0

7. Primary Outcome: Percentage of Participants Who Have Severe Hypoglycemia at Least Once Post-dose During Dosing For Part 1
Description: Severe hypoglycemia was defined as an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
Time Frame: Up to Day 20
Population: Safety Analysis Set included of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg | Part 1: Placebo Cohort 1-2
Number analyzed (Participants) | 6 | 6 | 4
percentage of participants | 0 | 0 | 0

8. Primary Outcome: Percentage of Participants Who Have Severe Hypoglycemia at Least Once Post-dose During Dosing For Part 2
Description: as for outcome 7
Time Frame: Up to Day 13
Population: Safety Analysis Set included of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg | Part 2: Placebo Cohort 1-4
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
percentage of participants | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Cmax: Maximum Plasma Concentration for TAK-648 for Part 1
Time Frame: Days 1 and 17 pre-dose and multiple time-points post-dose (Up to 72 hours)
Population: The Pharmacokinetic (PK) Set included all participants in the safety set with at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg
Number analyzed (Participants) | 6 | 6
ng/mL
  Day 1 | 6.342 (1.3552) | 16.150 (3.2073)
  Day 17 | 7.950 (2.3885) | 16.283 (4.6521)

10. Secondary Outcome: Cmax: Maximum Plasma Concentration for TAK-648 for Part 2
Time Frame: Days 1 and 10 pre-dose and multiple time-points post-dose (Up to 72 hours)
Population: The PK Set included all participants in the safety set with at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mg/mL
  Day 1 | 0.764 (0.2436) | 1.955 (0.3455) | 5.925 (1.9491) | 10.080 (5.2665)
  Day 10 | 0.670 (0.2054) | 2.355 (0.1499) | 6.430 (2.5774) | 9.612 (3.5611)

11. Secondary Outcome: Tmax: Time to Reach Maximum Plasma Concentration (Tmax) for TAK-648 for Part 1
Time Frame: Days 1 and 17 pre-dose and multiple time-points post-dose (Up to 72 hours)
Population: The PK Set included all participants in the safety set with at least 1 measurable plasma concentration.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg
Number analyzed (Participants) | 6 | 6
hours (hr)
  Day 1 | 0.500 [0.50 to 0.50] | 1.000 [0.50 to 1.50]
  Day 17 | 0.500 [0.50 to 1.00] | 0.710 [0.50 to 2.00]

12. Secondary Outcome: Tmax: Time to Reach Maximum Plasma Concentration (Tmax) for TAK-648 for Part 2
Time Frame: Days 1 and 10 pre-dose and multiple time-points post-dose (Up to 72 hours)
Population: The PK Set included all participants in the safety set with at least 1 measurable plasma concentration.
Measure: Median (Full Range); unit: hr
Arm/Group | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hr
  Day 1 | 1.000 [0.50 to 2.00] | 1.000 [0.50 to 1.50] | 1.000 [0.50 to 1.00] | 1.000 [0.50 to 1.50]
  Day 10 | 1.500 [1.00 to 2.00] | 0.750 [0.50 to 1.50] | 1.000 [0.50 to 1.50] | 1.000 [0.50 to 4.00]

13. Secondary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-648 for Part 1
Time Frame: Days 1 and 17 pre-dose and multiple time-points post-dose (Up to 72 hours)
Population: The PK Set included all participants in the safety set with at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg
Number analyzed (Participants) | 6 | 6
ng*hr/mL
  Day 1 | 31.676 (10.2111) | 88.168 (28.2484)
  Day 17 | 43.908 (18.4433) | 107.492 (39.6210)

14. Secondary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-648 for Part 2
Time Frame: Days 1 and 10 pre-dose and multiple time-points post-dose (Up to 72 hours)
Population: The PK Set included all participants in the safety set with at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL
  Day 1 | 5.018 (1.3681) | 14.861 (3.0267) | 38.878 (12.7876) | 63.376 (19.6130)
  Day 10 | 5.355 (1.5083) | 19.274 (3.5884) | 38.123 (14.0762) | 75.183 (35.8763)

15. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for TAK-648 for Part 1
Time Frame: Days 1 and 17 pre-dose and multiple time-points post-dose (Up to 72 hours)
Population: The PK Set included all participants in the safety set with at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg
Number analyzed (Participants) | 6 | 6
ng*hr/mL
  Day 1 | 31.973 (10.3893) | 89.043 (29.0630)
  Day 17 | 46.827 (21.8685) | 110.882 (41.8979)

16. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for TAK-648 for Part 2
Time Frame: Days 1 and 10 pre-dose and multiple time-points post-dose (Up to 72 hours)
Population: The PK Set included all participants in the safety set with at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL
  Day 1 | 5.147 (1.3861) | 15.078 (3.0768) | 39.160 (12.8099) | 64.694 (20.2316)
  Day 10 | 5.538 (1.5656) | 19.922 (3.8508) | 39.103 (14.5245) | 77.369 (36.7414)

17. Secondary Outcome: AUCtau: Area Under the Plasma Concentration-time Curve From Time 0 Over the Dosing Interval for TAK-648 for Part 1
Time Frame: Days 1 and 17 pre-dose and multiple time-points post-dose (Up to 72 hours)
Population: The PK Set included all participants in the safety set with at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg
Number analyzed (Participants) | 6 | 6
ng*hr/mL
  Day 1 | 30.209 (9.0944) | 82.148 (21.9186)
  Day 17 | 39.283 (15.7882) | 95.028 (28.9547)

18. Secondary Outcome: AUCtau: Area Under the Plasma Concentration-time Curve From Time 0 Over the Dosing Interval for TAK-648 for Part 2
Time Frame: Days 1 and 10 pre-dose and multiple time-points post-dose (Up to 72 hours)
Population: The PK Set included all participants in the safety set with at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL
  Day 1 | 4.833 (1.2018) | 13.902 (2.5432) | 36.570 (11.8662) | 59.507 (18.5291)
  Day 10 | 5.036 (1.3032) | 17.215 (2.8909) | 34.661 (13.0489) | 67.785 (28.2776)

ADVERSE EVENTS:
Time Frame: AEs were routinely collected from the time of first study drug administration until Follow-up Visit on Day 34 (±2) days (Part 1), and Day 26 (±2) days (Part 2).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1 Cohort 1: TAK-648 0.35 mg | Part 1 Cohort 2: TAK-648 0.80 mg | Part 1: Placebo Cohort 1-2 | Part 2 Cohort 1: TAK-648 0.05 mg | Part 2 Cohort 2: TAK-648 0.15 mg | Part 2 Cohort 3: TAK-648 0.35 mg | Part 2 Cohort 4: TAK-648 0.80 mg | Part 2: Placebo Cohort 1-4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 5/6 | 2/6 | 4/4 | 6/6 | 2/6 | 4/6 | 5/6 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1: TAK-648 0.35 mg (N=6) | Part 1 Cohort 2: TAK-648 0.80 mg (N=6) | Part 1: Placebo Cohort 1-2 (N=4) | Part 2 Cohort 1: TAK-648 0.05 mg (N=6) | Part 2 Cohort 2: TAK-648 0.15 mg (N=6) | Part 2 Cohort 3: TAK-648 0.35 mg (N=6) | Part 2 Cohort 4: TAK-648 0.80 mg (N=6) | Part 2: Placebo Cohort 1-4 (N=8)
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 2
Application site dermatitis (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Application site pruritus (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Application site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure orthostatic decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.